CLINICAL TRIAL: NCT07204704
Title: EUREKA: Evaluating Ultraviolet Radiation Exposure in Kids for Adaptive Intervention
Acronym: EUREKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCI121617
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUREKA Intervention (Other): This arm will utilize a SmartPhone app to deliver assessments and interventions for 21 days
  Interventions: Behavioral: EUREKA Intervention

INTERVENTIONS:
Behavioral: EUREKA Intervention — Participants will be asked to complete brief questionnaires about the child's sun protection up to six times daily throughout the study. During Week 2, participants will receive feedback and advice messages immediately after completing the questionnaires. During that week, participants will also be asked to collaboratively complete an action planning exercise (delivered to the child's phone) to plan sun protection for a selected outdoor activity that is likely to take place the next day.

SUMMARY:
This project will pilot a Just In Time Adaptive Intervention (JITAI) approach to providing feedback on child UVR exposure to children and their parents, with the ultimate goal of improving child use of sun protection strategies (e.g., use of sunscreen, protective clothing) and decreasing UVR exposure and sunburn occurrence. This study will utilize a SmartPhone app. If participants do not have a smartphone, they will be provided with one to use the app.

DETAILED DESCRIPTION:
Melanoma is the 6th most common form of cancer in the United States and its incidence has been increasing for the past three decades. While individuals diagnosed with melanoma have a generally optimistic prognosis (overall 5-year survival rates of 91%), once melanoma has metastasized to distant organs, the survival rate drops to only 17%. As a result, prevention and early detection of melanoma when it is more easily treated are of prime importance. Ultraviolet radiation (UVR) exposure is the primary modifiable risk factor for melanoma. Adoption of sun protective behaviors, such as sunscreen use, are essential for decreasing acute (sunburn) and long-term (DNA damage) effects of UVR exposure. Minimizing excess UVR exposure is especially important during childhood since childhood sunburns are a risk factor for melanoma.

Existing interventions for skin cancer prevention in childhood have not been able to provide children and families with real-time feedback and associated prompts related to the child's UVR exposure. Previous research has shown that families struggle with knowing how much UVR exposure their children obtain throughout the course of the day. JITAIs offer a unique opportunity to provide children and their parents with real-time feedback on the child's UVR exposure, as well as reminders for the child to use recommended sun protection strategies. Previous JITAIs have been observed to be effective at reducing sedentary activities, preventing relapse related to alcoholism, and helping with smoking cessation. However, JITAIs have been used more seldom among pediatric populations and have not yet been used to facilitate melanoma preventive strategies among children.

The overall goal of the proposed project is to pilot a JITAI approach to providing feedback on child UVR exposure to children and their parents, with the ultimate goal of improving child use of sun protection strategies (e.g., use of sunscreen, protective clothing) and decreasing UVR exposure and sunburn occurrence.

This study will utilize a SmartPhone app. Participants who provide informed consent and/or assent to participate in the study will be asked to complete activities on the app for 21 days. If children do not have a smartphone, they will be provided with one to use the app.

ELIGIBILITY:
Inclusion Criteria:

Parents:

* are at least 18 years old
* have at least one child between the ages of 8-17 who is living in the same household
* are the primary caregiver for the child participating in the study (defined as the individual who is responsible for daily implementation of health-related tasks for the child)
* have and are able to use a smartphone
* are willing to download and use a free smartphone app that will share their participating child's ultraviolet radiation exposure data with the research team.

Children:

* are 8 to 17 years old
* with a primary caretaker in Utah
* have no previous diagnosis of skin cancer
* have had a sunburn in the past year
* have used sunscreen and one other sun protection behavior never/rarely/sometimes in the past month (protective clothing items, shade when outdoors)
* are willing to wear a sensor (on their wrist or attached to their clothing) that collects data on ultraviolet radiation (UV) exposure

Exclusion Criteria:

Parents and Children:

* Do not speak, read/write English
* Have a pacemaker

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Self-reported child sun protection | From baseline to Post-Intervention, up to 21 days
  This outcome measure will report the frequency of self-report child sun protection using items that separately assess specific sun protection behaviors (e.g., sunscreen use).
Parent-reported child sun protection | From baseline to Post-Intervention, up to 21 days
  This outcome measure will report the frequency of parent-report child sun protection using items that separately assess specific sun protection behaviors (e.g., sunscreen use).

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Stump, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- University of Utah Department of Dermatology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Cancer Institute. SEER Stat Fact Sheets: Melanoma of the Skin. 2017; http://seer.cancer.gov/statfacts/html/melan.html.
- [Background] Armstrong BK, Kricker A. How much melanoma is caused by sun exposure? Melanoma Res. 1993 Dec;3(6):395-401. doi: 10.1097/00008390-199311000-00002. PMID 8161879
- [Background] Thomas JG, Bond DS. Behavioral response to a just-in-time adaptive intervention (JITAI) to reduce sedentary behavior in obese adults: Implications for JITAI optimization. Health Psychol. 2015 Dec;34S(0):1261-7. doi: 10.1037/hea0000304. PMID 26651467
- [Background] King AC, Hekler EB, Grieco LA, Winter SJ, Sheats JL, Buman MP, Banerjee B, Robinson TN, Cirimele J. Harnessing different motivational frames via mobile phones to promote daily physical activity and reduce sedentary behavior in aging adults. PLoS One. 2013 Apr 25;8(4):e62613. doi: 10.1371/journal.pone.0062613. Print 2013. PMID 23638127
- [Background] Free C, Knight R, Robertson S, Whittaker R, Edwards P, Zhou W, Rodgers A, Cairns J, Kenward MG, Roberts I. Smoking cessation support delivered via mobile phone text messaging (txt2stop): a single-blind, randomised trial. Lancet. 2011 Jul 2;378(9785):49-55. doi: 10.1016/S0140-6736(11)60701-0. PMID 21722952